CLINICAL TRIAL: NCT03482726
Title: Cadence Modulation to Improve Well-Being, Kinematics and Aerobic Performance in Cyclists
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2017-0131; A536110 (Other: UW Madison); SMPH\ORTHOPEDIC&REHAB\ORTHO (Other: UW Madison)
Record Dates: First submitted 2017-11-22; First posted 2018-03-29 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-04

CONDITIONS: Healthy
Keywords: bicycle; cadence; cyclist; modulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cycling Cadence Modulation (Other): 3 initial visits to collect baseline information; 6-week HIIT indoor cycling program at the individual prescribed cadence; final study visit for post-intervention measures.
  Interventions: Behavioral: Cycling Cadence Modulation

INTERVENTIONS:
Behavioral: Cycling Cadence Modulation — 6-week high intensity training (HIIT) indoor cycling program, described later, at their prescribed cadence (FCC or EOC), using cadence meters.

SUMMARY:
This study will utilize a combination of cardiovascular analysis, 3D motion capture, and a software package, Metrifit, to monitor measures of well-being to comprehensively evaluate both the musculoskeletal and physiological responses following a HIIT training intervention at EOC as a means of improving performance and potentially reducing injury risk factors. This holistic approach of physiological and biomechanical factors is unprecedented. This is the first interventional study to determine the effect of high intensity training at EOC on cardiovascular performance, kinematics and well-being which may minimize risk of injury factors.

DETAILED DESCRIPTION:
In the first session, each individual will be asked to fill out a questionnaire to regarding cycling experience, prior bike fits (with data sheets when available), and injury history. Maximal aerobic capacity (VO2max) will be determined. During the test, subjects will be asked rate exertion. Before testing, the system will be calibrated with known oxygen and carbon dioxide concentrations. During the test, subjects will be asked to breathe normally through a low dead space bidirectional turbine. Inspired and expired gases will be analyzed for concentrations of O2 and CO2, to determine alveolar gas exchange. Total ventilation (VE), respiratory rate, oxygen consumption (VO2), carbon dioxide (VCO2) will be measured, and respiratory exchange ratio (RER; VCO2/VO2) will be calculated continuously during the test and expressed as a 30-second rolling average.

Participants will return 48 hours later, at which time EOC will be determined after a moderate intensity prolonged cycling exercise (PCE) at seven different cadences. Cadences from 50rpm to 110rpm will be randomly generated and introduced every 3 minutes, followed by a 3 minute cool down at FCC at 40% PP (Figure Subjects will then be pair matched by gender and randomized into control (FCC) or EOC modulation groups.

48 hours following EOC testing, subject will return for a second progressive maximal cycling test performed at FCC or EOC based on group assignment.

Subjects will then participate in a 6 week high intensity training (HIIT) indoor cycling program at their prescribed cadence (FCC or EOC), using cadence meters. Training will consist of three non-consecutive days each week for 60 min, and alternate between two HIIT workouts. Resistance will be increased to meet the HIIT requirement, while cadence will remain at FCC or EOC. Subjects will be asked to warm-up at a light (3/10) workload for 10 minutes, followed by HIIT consisting of 4 minutes at an intensity of 8/10 on the modified Borg, and 90 seconds recovery (2/10). This will be repeated 8 times, followed by 10 minutes of cool down. The alternating HIIT workout will include a 10 minute warm up, followed by 12 intervals lasting 2 minutes at an RPE of 9/10 and 3 minutes of recovery. The session will conclude with a 10 minute cool down.

Within one week of completing their training program, subjects will return for their fourth and final study visit, at which time a VO2max test and kinematic data collection will be repeated at FCC or EOC.

ELIGIBILITY:
Inclusion Criteria:

1. An experienced cyclist will be defined as one with at least 5 years of cycling experience and 5000 miles of training on a road bike with a clipless pedal system.
2. Able to tolerate strenuous, maximal exercise and comply with a 6 week training protocol
3. Have access to an indoor trainer or spin bike with a cadence sensor in order to train 3 times per week for 60 minutes

Exclusion Criteria:

1. Taking medication which could impact cardiovascular function or performance (stimulants, beta-blockers, e.g.)
2. Significant cardiac or pulmonary disease (congenital cardiac disease, uncontrolled hypertension, uncontrolled asthma, e.g.)
3. Musculoskeletal injuries that preclude a maximal cycling effort and participation in training program

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Time to exhaustion T(max) | Baseline
  time to reach exhaustion
Ventilatory threshold (VT) | Baseline
Maximal cardiac output | Baseline
Maximal stroke volume | Baseline
decreased trunk lean | Baseline
  decrease in degree of lean in truck
decreased ankle dorsiflexion | Baseline
  decrease in amount of ankle dorsiflexion
decreased knee splay | Baseline
  decreased degree of knee splay

SECONDARY OUTCOMES:
Improved VO2 max | 6 weeks
  Increased maximum O2 volume
Increased O2 consumption at VT | 6 weeks
  Improved oxygen consumption at ventilatory threshold
Time to VT | 6 weeks
  Improved time to reach ventilatory threshold
Time to T(max) | 6 weeks
  Improved time to reach exhaustion
decreased trunk lean | 6 weeks
  decrease in degree of lean in truck
decreased ankle dorsiflexion | 6 weeks
  decrease in amount of ankle dorsiflexion
decreased knee splay | 6 weeks
  decreased degree of knee splay
change in overall soreness and fatigue | 6 weeks
  decrease in reported soreness and fatigue as measured and reported via Metrifit software

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Watson, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States